CLINICAL TRIAL: NCT00178139
Title: Music Therapy as an Adjunctive Treatment in the Management of Stress for Patients Being Weaned From Mechanical Ventilation
Brief Title: Music Therapy for Patients Being Weaned From Mechanical Ventilation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Arthur Flager Fultz Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10243
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Insufficiency
Keywords: Music Therapy; Mechanical ventilation; Weaning from mechanical ventilation; complementary and alternative therapy
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Music Therapy — Music Therapy

SUMMARY:
The purpose of the study is to determine whether Music Therapy interventions can be used as supportive therapy for patients undergoing weaning from mechanical ventilation. The music will support the procedure by serving as a stimulus for relaxation and/or pain and anxiety management.Music used is varied according to subject's preferences.

DETAILED DESCRIPTION:
Music therapy interventions will be used as supportive therapy for patients undergoing weaning from mechanical ventilation. The music will support the procedure by serving as a stimulus for relaxation and/or pain and anxiety management. The intervention will consist of 40 - 50 minutes of active music therapy and improvisation in which the music is used as a distraction from the hospital setting and the procedure taking place. The intervention will end with 5 to 10 minutes of discussion of music activities/selections to be used between music therapy sessions. The intervention is individualized and can be modified accordingly to the subject's preferences.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety
* weaning sessions less than 8 hours

Exclusion Criteria:

weaning trials greater than 8 hours

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of music therapy interventions in assisting patient to be liberated from mechanical ventilation more quickly than control subjects. | prospective

SECONDARY OUTCOMES:
Exploratory hypotheses will investigate decreased anxiety measured by -physiologic measures | prospective
- decreased use of anxiolytic, antidepressant and antipsychotic agents. | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Olle Jane Z Sahler, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Result] Oliva R, Hunter BC, Sahler OJZ, Gaisser D, Salipante DM. (2009). The Use of Music Therapy for Patients Being Weaned from Mechanical Ventilation: A Pilot Study. In Azoulay R & Loewy J (eds). Music, the Breath and Health: Advances in Integrative Music Therapy. New York: Satchnote Press.